CLINICAL TRIAL: NCT05780983
Title: Sleep Well 24 (SWELL24): Promoting Healthy Sleep-wake Behaviors Across a 24-hour Cycle in Frail Older Adults
Brief Title: Sleep Well 24 (SWELL24) Healthy Sleep-Wake Behaviors in Older Adults
Acronym: SWELL24
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00089122; P30AG021332 (NIH)
Record Dates: First submitted 2023-03-10; First posted 2023-03-23 (Actual); Results first posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-01

CONDITIONS: Insomnia Disorder
Keywords: sleep-wake patterns; poor sleep
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: All participants enrolled in the pilot trial will receive the intervention, all activities will be unblinded. Older adults utilizing outpatient primary care clinics belonging Atrium Wake Forest Baptist Health. All activities will take place within a clinical setting. Participants will be asked to monitor their sleep-activity behaviors while at home.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- education and coaching on developing healthy nighttime sleep and daytime activity behaviors (Other): The intervention includes a four-session, in-person program delivered by a Master's-level provider. Each individual session will be approximately 30-45 minutes in length. Each session will include education and coaching on developing healthy nighttime sleep and daytime activity behaviors.
  Interventions: Behavioral: education and coaching on developing healthy nighttime sleep and daytime activity behaviors

INTERVENTIONS:
Behavioral: education and coaching on developing healthy nighttime sleep and daytime activity behaviors — The intervention includes a four-session, in-person program delivered by a Master's-level provider. Each individual session will be approximately 30-45 minutes in length. Each session will include education and coaching on developing healthy nighttime sleep and daytime activity behaviors.

SUMMARY:
To finalize daytime intervention components for a comprehensive sleep-wake intervention for frail older adults and explore feasibility and acceptability using a pilot trial.

DETAILED DESCRIPTION:
An enhanced intervention addressing both nighttime and daytime activities will be developed based on prior evidence and further informed by data. A successive cohort design will be utilized to evaluate and refine key intervention components and gather feedback on older adults' experiences.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or over
* One or more outpatient primary care visits to Wake Forest Baptist Health in the prior 12 months
* Meets diagnostic criteria for Insomnia Disorder
* Less than 30 minutes of daily activity or less than 150 minutes total weekly activity for one month or longer, as reported on brief telephone screener
* Able to ambulate safely (with or without an assistive device)
* Able to follow study directions
* Able to communicate and follow study instructions
* English speaking

Exclusion Criteria:

* Untreated organic sleep disorder (e.g., central or obstructive sleep apnea, restless leg syndrome)
* Serious or unstable medical or psychiatric condition that would prevent participation in a behavioral intervention (e.g., terminal illness, uncontrolled psychiatric disorder, substance abuse disorder)
* Lack of decision-making capacity, as documented in medical record
* Referred to institutional care and/or currently residing in a nursing home or other residential facility

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 7 (Actual)
Dates: Start 2024-05-08 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaime M Hughes, PhD, MPH, MSW, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Education and Coaching on Developing Healthy Nighttime Sleep and Daytime Activity Behaviors
Started | 7
Completed | 6
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Education and Coaching on Developing Healthy Nighttime Sleep and Daytime Activity Behaviors
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Education [Mean (Full Range); unit: years] | 14.9 [10 to 18]

OUTCOME MEASURES:

1. Primary Outcome: Sleep Efficiency
Description: Total number of minutes asleep divided by total time in bed measure by wrist actigraph
Time Frame: Month 2
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Education and Coaching on Developing Healthy Nighttime Sleep and Daytime Activity Behaviors
Number analyzed (Participants) | 6
percent | 95.1 (1.7)

2. Secondary Outcome: Insomnia Severity Scores
Description: Insomnia Severity Index (ISI) is a 7-item validated, self-report questionnaire used to evaluate insomnia severity. Scores range from 0 - 28, higher scores indicate more severe insomnia symptom severity.
Time Frame: Month 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Education and Coaching on Developing Healthy Nighttime Sleep and Daytime Activity Behaviors
Number analyzed (Participants) | 6
score on a scale | 9.67 (9.7)

3. Secondary Outcome: Total Daytime Activity
Description: Daily activity (total count of steps), per wrist actigraph
Time Frame: Month 2
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Education and Coaching on Developing Healthy Nighttime Sleep and Daytime Activity Behaviors
Number analyzed (Participants) | 6
steps | 5188 (2475)

4. Secondary Outcome: Pittsburgh Sleep Quality Index Score
Description: Pittsburgh Sleep Quality Index: Daily Disturbances score using the 3-factor scoring model, per self-reported assessment. Scores range from 0-6. Higher scores indicate more daily disturbance.
Time Frame: Month 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Education and Coaching on Developing Healthy Nighttime Sleep and Daytime Activity Behaviors
Number analyzed (Participants) | 6
score on a scale | 1.2 (0.4)

ADVERSE EVENTS:
Time Frame: Baseline through post-program assessment (month 2)
Arm/Group | Education and Coaching on Developing Healthy Nighttime Sleep and Daytime Activity Behaviors
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2024-05-02): https://cdn.clinicaltrials.gov/large-docs/83/NCT05780983/Prot_001.pdf
  • Statistical Analysis Plan (2025-10-17): https://cdn.clinicaltrials.gov/large-docs/83/NCT05780983/SAP_002.pdf
  • Informed Consent Form (2024-05-07): https://cdn.clinicaltrials.gov/large-docs/83/NCT05780983/ICF_000.pdf